CLINICAL TRIAL: NCT06065527
Title: Future Planning and Well-Being for Individuals With Intellectual Disabilities and Family Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Baylor College of Medicine (Other); Christiana Care Health Services (Other); Children's Hospital of Philadelphia (Other); Children's Hospital Medical Center, Cincinnati (Other); Geisinger Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-0381
Record Dates: First submitted 2023-09-26; First posted 2023-10-04 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Intellectual Disability
Keywords: Caregiver; case management
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Intervention Model Description: This is a multi-site, two-arm, pragmatic randomized controlled trial (RCT) of primary family caregivers of individuals with IDD. Family caregivers will be randomized 1:1 to one of 2 treatment arms described above. This is a non-blinded study because the nature of the intervention prevents participants from being blinded to their study arm.
Masking Description: Masking will not occur because it is not a blinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced usual care and Map Our Life (Active Comparator): Participants will be introduced to Map Our Life, by research staff. In accordance to the Preparation for Future Care Model, PYL: (1) introduces users to long-term care (LTC) related choices (care expectation); (2) assesses the unique caregiving needs of the care recipient (awareness); (3) educates the users on locally and nationally available home-based resources (information gathering); (4) makes choices about LTC preferences (decision-making), and (5) shares those choices with others (concrete planning).This process is associated with informed and value-based decisions that fit the preferences of the care recipient and increased well-being according to the theory of proactive coping, which states that preparation for future stressors improves the ability to cope in real-time.
  Interventions: Behavioral: Map Our Life
- Enhanced usual care and Attention Control (Placebo Comparator): In this arm, caregivers will be referred to a website containing information from "Disability and Health Information for Family Caregivers". The content in the attention control is from CDC-sponsored websites that promote healthy activities and behaviors targeting people with disabilities and their family caregivers. Additionally, the content leads users to CDC-sponsored "Caregiving" webpages which assist families in developing care plans. All content is available in English and Spanish.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Map Our Life — The intervention takes participants through the process of planning using the Preparation for Future Care Model stages: care expectation, awareness, information gathering, decision making, and concrete planning. The intervention has 8 modules: (1) Letter of Intent for Your Loved One, (2) Caregiver Support and Well-Being, (3) Medical Decision Making for Your Loved One, (4) Daily Routines and Medical Management, (5) Medicaid Waiver for Your Loved One, (6) Financial Planning for Your Loved One, (7) Emergency Planning for Your Loved One, and (8) Managing Jobs, Day Programs, and Transportation. Map Our Life takes users - the caregiver alongside the individual with intellectual disability - through the stages of planning in each of the 8 modules until a concrete care plan is developed. The last component of the intervention is that this Care Plan is subsequently saved and shared with others such as care managers, clinicians, friends or family members.
  Arms: Enhanced usual care and Map Our Life
Behavioral: Attention Control — The control group will have access to a CDC Website, CDC Healthy Living with a Disability.
  Arms: Enhanced usual care and Attention Control

SUMMARY:
This study will compare the effectiveness of a web-based long-term care planning tool (Map Our Life) partnered with traditional case management services to traditional case management services partnered with an attention-control Centers for Disease Control and Prevention (CDC) sponsored website on health promotion for people with disabilities. The goal of this clinical trial is to promote long-term care (LTC) knowledge and planning among individuals with intellectual/developmental disabilities (IDD) and their family caregivers to improve social supports, health, and quality of life outcomes.

DETAILED DESCRIPTION:
People with intellectual/developmental disabilities (IDD) experience alarmingly high rates of mortality, morbidity, and acute care utilization compared to those without an IDD, particularly during emergencies. Caregiver health and well-being is a determinant of health outcomes for people with an IDD. Yet, caregivers are aging and frequently experience high caregiver burden and poor well-being. Poor preparedness and planning lead to crises and harm, including emotional trauma, unsafe living conditions, unwanted emergent nursing home placements, and potential early mortality, for both people with an IDD and their family caregivers.

The goal of this study is to promote health emergency preparedness and long-term care (LTC) decision-making among individuals with intellectual/developmental disabilities (IDD) and their family caregivers to improve patient- and caregiver-reported health and quality of life outcomes. Through partnerships with adults with IDD, their families, IDD community organizations, and IDD services agencies, the investigators seek to conduct a randomized controlled trial comparing the effectiveness of Map Our Life - a web-based future planning intervention and enhanced usual care (EUC) - care coordination services vs. an attention control (AC) and EUC on health promotion for people with disabilities and their family caregivers. Aim 1 will compare the effectiveness of Map Our Life +EUC vs AC+EUC on family caregiver support and well-being at 1, 6, and 18 months. Aim 2 will examine the comparative effectiveness of Map Our Life +EUC vs. AC+EUC on planning behaviors and communicating future preferences for LTC planning, and its mediating effects on family caregiver support and well-being at 1, 6, and 18 months. Finally, aim 3 will identify how individual and caregiver need factors and access to services and supports moderate intervention treatment effects at 6 and 18 months from the perspective of the individual with IDD and separately from their caregiver.

We will conduct a national, multi-site, two-arm, randomized controlled trial (RCT) of primary family caregivers of individuals with IDD. A total of 1050 family caregivers will be randomized 1:1 to one of 2 treatment arms: (1) enhanced usual care plus a web-based future planning intervention, Map Our Life; and (2) attention control website plus EUC. Primary participants will be family caregivers of individuals with IDD who are at least 18 years old living in community settings recruited from stakeholder groups, Northwell Health (New York), Christiana Care Health System (Delaware), Baylor College of Medicine (Texas), Children's Hospital of Philadelphia (Pennsylvania), Cincinnati Children's Hospital Medical Center (Ohio), and Geisinger Health (Pennsylvania). Primary outcomes include caregiver burden and caregiver wellbeing. Secondary outcomes include adequacy and satisfaction with services and supports, well-being and planning choices of adult care recipient with IDD, and planning behaviors and communication of plans. Participants will complete surveys at the time of enrollment and at 1-, 6-, and 18- months post enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers of individuals with intellectual and/or developmental disabilities living in a community setting
* Ability to speak English or Spanish
* Access to a tablet, computer, or smartphone

Exclusion Criteria:

* Speaks a language other than English or Spanish
* Does not have access to a tablet, computer, or smartphone
* Caregivers who care for individuals with intellectual and developmental disabilities who are less than 10 years of age.
* Special populations such as: fetuses, prisoners, or other institutionalized individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Outcomes - Caregiver burden | Baseline, 1 month, 6 months and 18 months.
  The primary outcome measure is caregiver burden as measured by the Zarit Burden Interview (ZBI). The ZBI is the most commonly used measure of distress among caregivers, and has good clinimetric properties and responsiveness. Responses to each item in the scale are on a 5-point scale ranging from 0 ("Never") to 4("Nearly Always"), with a total score ranging from 0 to 88.

SECONDARY OUTCOMES:
Quality of Life Outcomes - Caregiver self-efficacy | Baseline, 1 month, 6 months and 18 months.
  The second outcome measure is self-efficacy as measured by the 5-item Respite Subscale of the Revised Scale for Caregiving Self-Efficacy, which has strong clinimetric properties and responsiveness. All questions start with the stem, "How confident are you that you can ask a friend or family member to stay with your loved one for…". An example is, "...a day when you need to see the doctor yourself?". Items are scored from 0 ("Cannot do at all") to 100 ("Certain can do"), for a total mean score ranging from 0 to 100.
Quality of Life Outcomes - IDD | Baseline and 6 months
  As part of an exploratory aim, the study will measure quality of life outcomes among affected individuals with intellectual disability using the World Health Organization Quality of Life Scale - Disability Modules (WHOQOL-Dis), a cross-cultural, multi-center instrument developed by the WHOQOL group for the assessment of quality of life in persons with disabilities. The scale was selected for its combination of specificity and validity among people with IDD and for its brevity and convenience.
Health Behaviors Outcomes - Problem-focused coping behaviors | Baseline, 1 month,6 months and 18 months.
  This outcome is problem-focused coping behaviors, as measured by the 4-item active coping, 4-item planning, 4-item seeking of instrumental social support, and 4-item denial subscales of the Coping Orientation to Problems Experienced (COPE) inventory, a multi-dimensional coping inventory to assess responses to stress. Items ask participants what they usually do when confronting difficult or stressful events in their lives, and include statements such as "I make a plan of action".
Health Behaviors Outcomes - Caregiver long term care planning behaviors | Baseline, 1 month,6 months and 18 months.
  This outcome focuses on long term care planning behaviors. This measure is adapted from the planning behaviors and communication of plans questionnaire used in the Plan Your Lifespan (PYL) randomized clinical trial of aging adults. Respondents answer on a 5-point Likert scale ranging from 1 ("Strongly disagree") to 5 ("Strongly agree"). Responses are summed creating a score ranging from 21 to 105, with higher scores indicating better planning and communication behavior.
Health Behaviors Outcomes - Caregiver long term care knowledge | Baseline, 1 month, 6 months, and 18 months
  This exploratory outcome will measure long term care knowledge, an enabling factor, measure by the Information and Planning Subdomain of the National Core Indicators (NCI) Family Surveys. Responses range from "Never" to "Always" and are summed based on the "Always" response.

CONTACTS AND LOCATIONS:
Locations (1):
- Cohen Children's Medical Center, New Hyde Park, New York, United States

REFERENCES:
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Schreiner AS, Morimoto T, Arai Y, Zarit S. Assessing family caregiver's mental health using a statistically derived cut-off score for the Zarit Burden Interview. Aging Ment Health. 2006 Mar;10(2):107-11. doi: 10.1080/13607860500312142. PMID 16517485
- [Background] Lindquist LA, Ramirez-Zohfeld V, Sunkara PD, Forcucci C, Campbell DS, Mitzen P, Ciolino JD, Gregory D, Kricke G, Cameron KA. PlanYourLifeSpan.org - an intervention to help seniors make choices for their fourth quarter of life: Results from the randomized clinical trial. Patient Educ Couns. 2017 Nov;100(11):1996-2004. doi: 10.1016/j.pec.2017.06.028. Epub 2017 Jun 27. PMID 28689855
- [Background] Lindquist LA, Ramirez-Zohfeld V, Sunkara PD, Forcucci C, Campbell DS, Mitzen P, Ciolino JD, Kricke G, Seltzer A, Ramirez AV, Cameron KA. Helping Seniors Plan for Posthospital Discharge Needs Before a Hospitalization Occurs: Results from the Randomized Control Trial of PlanYourLifespan.org. J Hosp Med. 2017 Nov;12(11):911-917. doi: 10.12788/jhm.2798. Epub 2017 Aug 23. PMID 29091979
- [Background] Ramirez-Zohfeld V, Seltzer A, Ramirez A, Muhammad R, Lindquist LA. Longitudinal Follow-Up of Long-Term Care Planning Using PlanYourLifespan.org. J Appl Gerontol. 2021 May;40(5):536-540. doi: 10.1177/0733464820943066. Epub 2020 Jul 19. PMID 32686545
- [Background] Rydzewska E, Hughes-McCormack LA, Gillberg C, Henderson A, MacIntyre C, Rintoul J, Cooper SA. Prevalence of long-term health conditions in adults with autism: observational study of a whole country population. BMJ Open. 2018 Sep 1;8(8):e023945. doi: 10.1136/bmjopen-2018-023945. PMID 30173164
- [Background] Kinnear D, Morrison J, Allan L, Henderson A, Smiley E, Cooper SA. Prevalence of physical conditions and multimorbidity in a cohort of adults with intellectual disabilities with and without Down syndrome: cross-sectional study. BMJ Open. 2018 Feb 5;8(2):e018292. doi: 10.1136/bmjopen-2017-018292. PMID 29431619
- [Background] Indicators | National Core Indicators. Accessed April 30, 2020. https://www.nationalcoreindicators.org/about/indicators/
- [Background] CDC. Disability & Health Information for Family Caregivers | CDC. Centers for Disease Control and Prevention. Published October 28, 2019. Accessed January 11, 2022. https://www.cdc.gov/ncbddd/disabilityandhealth/family.html
- [Background] Power MJ, Green AM; WHOQOL-Dis Group. Development of the WHOQOL disabilities module. Qual Life Res. 2010 May;19(4):571-84. doi: 10.1007/s11136-010-9616-6. Epub 2010 Mar 9. PMID 20217246
- [Derived] Steinway C, Wright C, Kwak S, Teng O, Seide A, Berens J, Woodward J, Riddle I, Davis T, Greenberg A, Szalda D, Shults J, Cerise J, Jan S. Innovative Web-Based Future Planning and Well-Being for Caregivers of Individuals With Intellectual and Developmental Disabilities: Protocol of a Pragmatic Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 1;14:e77184. doi: 10.2196/77184. PMID 41032360